CLINICAL TRIAL: NCT07257523
Title: Carbon Ion Radiotherapy in Frail Patients With Pancreatic Cancer: A Prospective Phase II Study
Brief Title: Carbon Ion Radiotherapy in Frail Patients With Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2025-0681
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Intervention Model Description: This study is a prospective, single-arm phase II clinical trial evaluating the efficacy and safety of carbon ion radiotherapy in frail patients with non-metastatic pancreatic cancer who are not eligible for surgery or systemic chemotherapy.
Masking Description: This is an open-label study with no blinding. All participants and investigators are aware of the assigned intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carbon Ion Radiotherapy (Experimental): Participants receive carbon ion radiotherapy delivered either as 55.2 Gy in 12 fractions over 3 weeks or 40-48 Gy in 4 fractions over 1 week. Treatment planning includes 4D-CT-based simulation, defined target volumes (GTV/CTV), and organ-at-risk dose constraints. Radiotherapy is administered with daily or alternate-day fractionation depending on the selected regimen.
  Interventions: Other: Carbon Ion Radiotherapy

INTERVENTIONS:
Other: Carbon Ion Radiotherapy — Carbon ion radiotherapy is delivered with two possible regimens: 55.2 Gy in 12 fractions over 3 weeks or 40-48 Gy in 4 fractions over 1 week. Treatment planning is performed using contrast-enhanced CT and 4D-CT to assess respiratory motion. Target volumes include the gross tumor volume and high-risk peripancreatic regions, while organs at risk (stomach, duodenum, bowel, liver, kidneys, spinal cord) follow strict dose constraints. Treatments are delivered once daily for the 12-fraction regimen or on alternate days for the 4-fraction regimen. Adaptive planning may be applied if weekly evaluation CT identifies anatomic changes. Acute and late toxicities are monitored throughout treatment using CTCAE v5.0.

SUMMARY:
"This prospective, single-arm phase II study aims to evaluate the efficacy and safety of carbon ion radiotherapy in frail patients with histologically confirmed, non-metastatic pancreatic cancer who are not eligible for surgery or systemic chemotherapy. Frail status is defined as a Clinical Frailty Scale (CFS) score ≥4 or the presence of significant medical comorbidities limiting aggressive treatment.

Carbon ion radiotherapy, known for its superior dose distribution and high linear energy transfer, may offer improved tumor control with acceptable toxicity in this vulnerable population. This study will assess overall survival, progression-free survival, local control, toxicity, and quality of life.

DETAILED DESCRIPTION:
"This prospective, single-arm phase II study evaluates the efficacy and safety of carbon ion radiotherapy in frail patients with non-metastatic pancreatic cancer who are not eligible for surgery or systemic chemotherapy due to a Clinical Frailty Scale (CFS) score ≥4 or significant medical comorbidities. carbon ion radiotherapy provides superior dose distribution and higher biological effectiveness compared with conventional X-ray radiotherapy, offering a potentially effective treatment option for this clinically vulnerable population.

Participants will undergo baseline evaluations including imaging (CT/MRI/PET-CT), laboratory tests, tumor markers, frailty assessment, and quality-of-life questionnaires (EORTC QLQ-C30 and FACT-Hep). Carbon ion radiotherapy will be delivered using 4D-CT-based planning, with either 55.2 Gy (RBE) in 12 fractions or 40-48 Gy (RBE) in 4 fractions. Target volumes include the primary tumor and high-risk peripancreatic regions, while organs-at-risk such as the stomach, duodenum, bowel, liver, kidneys, and spinal cord follow strict dose constraints. Weekly on-treatment assessments will monitor acute toxicity using CTCAE v5.0, and adaptive planning will be performed if needed.

Post-treatment follow-up will occur at 1-3 months and every 3-6 months thereafter for up to 2 years, including imaging, toxicity evaluation, tumor marker assessment, and repeated QOL surveys.

The primary endpoint is overall survival. Secondary endpoints include progression-free survival, local control, treatment-related toxicity, quality of life, and tumor marker changes. Survival analyses will use Kaplan-Meier and Cox regression methods, and quality-of-life and toxicity outcomes will be summarized descriptively.

ELIGIBILITY:
Inclusion Criteria:

- Histologically confirmed pancreatic cancer without distant metastasis.

Not eligible for surgery or systemic chemotherapy, defined as:

Clinical Frailty Scale (CFS) score ≥ 4, or Significant medical comorbidities precluding standard treatment. Patients who decline surgery and chemotherapy after adequate counseling. Age ≥ 19 years. Able to provide written informed consent. Eligible and willing to receive carbon ion radiotherapy.

Exclusion Criteria:

* Age < 19 years. Presence of distant metastasis at baseline imaging (CT/MRI/PET-CT). Active or uncontrolled infection that may interfere with treatment. Active bleeding or bleeding tendency requiring immediate medical intervention. Pregnant or breastfeeding women. Any condition that, in the investigator's judgment, makes participation unsafe or inappropriate (e.g., severe organ dysfunction preventing radiotherapy).

Inability to comply with study procedures or follow-up schedule.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival in frail patients with pancreatic cancer receiving carbon ion radiotherapy | Up to 2 years from the start of treatment
  Overall survival will be assessed from the date of treatment initiation to death from any cause. The study will determine whether carbon ion radiotherapy provides a clinically meaningful improvement in survival compared with historical outcomes in frail patients with pancreatic cancer who previously received only supportive care or conventional X-ray radiotherapy.

SECONDARY OUTCOMES:
Progression-free survival | Up to 2 years from the start of treatment
  Progression-free survival will be measured from the start of carbon ion radiotherapy to radiologic tumor progression or death from any cause, whichever occurs first.
Local control rate | Up to 2 years from the start of treatment
  Local control will be assessed through serial CT, MRI, or PET-CT imaging to determine the absence of local tumor progression within the irradiated region.
Quality of Life: EORTC QLQ-C30 Score | Baseline, end of radiotherapy, and every 3-6 months up to 2 years
  Quality of life will be assessed using the EORTC QLQ-C30 questionnaire. The score ranges from 0 to 100. Higher scores indicate a higher response level (or better functioning/worse symptom, depending on the scale).
Treatment-related toxicity | During radiotherapy and every 3-6 months up to 2 years
  Acute and late toxicities will be recorded and graded according to CTCAE version 5.0 to evaluate the safety profile of carbon ion radiotherapy in frail pancreatic cancer patients.
Tumor marker changes (CA 19-9, CEA) | Baseline and every follow-up visit up to 2 years
  Changes in tumor markers (CA 19-9 and CEA) will be monitored to assess treatment response trends following carbon ion radiotherapy.
Quality of Life: FACT-Hep Score | Baseline, end of radiotherapy, and every 3-6 months up to 2 years
  Secondary Outcome - Quality of life will be assessed using the FACT-Hep questionnaire. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No